CLINICAL TRIAL: NCT00991588
Title: Reconstruction of the Posterior Cruciate Ligament and Posterolateral Structures of the Knee
Brief Title: Clinical Outcome of Posterior Cruciate Ligament (PCL) Posterolateral Reconstruction
Status: Completed | Type: Observational
Sponsor: Sue Barber-Westin (Other)
Responsible Party: Sponsor-Investigator, Sue Barber-Westin, Director Clinical Studies, Cincinnati Sportsmedicine Research and Education Foundation
Organization: Cincinnati Sportsmedicine Research and Education Foundation (Other)
Other Study IDs: PCLPL-001
Record Dates: First submitted 2009-10-06; First posted 2009-10-08 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Knee Injuries
Keywords: PCL; Posterolateral
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PCL, posterolateral reconstruction: All patients who are entered into study who receive a PCL and/or posterolateral knee ligament reconstruction
  Interventions: Procedure: PCL, posterolateral reconstruction

INTERVENTIONS:
Procedure: PCL, posterolateral reconstruction — The operative procedures involve either a single- or double-strand PCL graft which is usually harvested from the patient's knee. In cases of multiple ligament procedures, allograft tissues may be used which are obtained from tissue banks certified by the American Associate of Tissue Banks and that have passed FDA inspection. The posterolateral structures, including the fibular collateral ligament (FCL), are reconstructed with one or two grafts, depending upon the severity of damage encountered at surgery.

SUMMARY:
The purpose of this investigation is to determine the clinical outcome of surgical reconstruction of complete ruptures to the posterior cruciate ligament (PCL) and posterolateral structures of the knee joint. The outcome will be determined with validated and rigorous knee rating systems between 2 and 10 years postoperatively. The results will be determined by the analysis of subjective and functional factors, sports and occupational activity levels, a comprehensive physical examination, and a radiographic evaluation. We hypothesize that the appropriately indicated procedures will effectively restore normal knee stability and function in patients with isolated or combined injuries to these structures.

DETAILED DESCRIPTION:
Because injuries to the PCL and posterolateral structures occur with less frequency than other structures in the knee joint (such as the anterior cruciate ligament and menisci), fewer studies are available to assist the surgeon and patient with appropriate decision-making regarding conservative versus surgical treatment. The majority of patients who sustain injury to these structures are treated conservatively. Unfortunately, several investigations describe noteworthy symptoms and functional limitations following conservative management, and a high percentage of patients develop knee osteoarthritis that can be disabling for both recreational and daily activities. The investigators of this study have nearly three decades of experience and have extensively studied the effects of this injury in both the laboratory and clinic settings. It is our opinion that surgical reconstruction provides significant benefit when appropriately indicated, as has been demonstrated in our previous studies. Especially in athletic individuals, PCL and posterolateral reconstructive procedures have advanced to the point where more predictable results can be expected to restore sufficient knee function. Studies have demonstrated, at least in the short-term, that the majority of patients with acute ligament ruptures treated with reconstruction are able to return to various levels of sports activities.12 Whether these procedures will decrease the risk of the patient developing future osteoarthritis is unknown and requires further study.

ELIGIBILITY:
Inclusion Criteria:

* Complete rupture to the posterior cruciate ligament, greater than 10 mm of increased posterior tibial translation
* Rupture to the posterolateral knee structures, greater than 5 mm of increased lateral tibiofemoral joint opening, greater than 10 degrees of increased external tibial rotation
* Patient willing to comply with postoperative rehabilitation program

Exclusion Criteria:

* Patient unwilling to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled for PCL and/or posterolateral reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Elimination of knee giving-way | Minimum 2 years postoperatively

SECONDARY OUTCOMES:
Posterior tibial translation | Minimum 2 years postoperative
Lateral tibiofemoral joint opening | Minimum 2 years postoperatively
External tibial rotation | Minimum 2 years postoperatively
Elimination of knee pain | Minimum 2 years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Frank Noyes, M.D., Principal Investigator — Cincinnati Sportsmedicine Research and Education Foundation
Locations (1):
- Cincinnati Sportsmedicine and Orthopaedic Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes